CLINICAL TRIAL: NCT03373487
Title: Cognitive Rehabilitation in Brain Tumor Patients After Neurosurgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Elisabeth-TweeSteden Ziekenhuis (Other)
Collaborators: Tilburg University (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other); Erasmus Medical Center (Other); Medical Center Haaglanden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 842003009
Record Dates: First submitted 2017-09-05; First posted 2017-12-14 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2017-10

CONDITIONS: Brain Tumor, Primary; Cognitive Impairment
MeSH Terms: conditions — Brain Neoplasms; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Well-trained research assistants, who are conducting neuropsychological assessments, are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early-intervention group (Experimental): Patients follow the evidence-based cognitive rehabilitation program ReMind, which is provided via an iPad. It incorporates psychoeducation, strategy training and retraining. The intervention commenced 3 months after surgery and patients were advised to spend 3 hours per week on the program for 10 weeks.
  Interventions: Behavioral: The cognitive rehabilitation program ReMind
- Waiting-list control group (Other): The waiting-list control group will be offered the same cognitive rehabilitation program after they have undergone all study assessments one year after surgery.
  Interventions: Behavioral: The cognitive rehabilitation program ReMind

INTERVENTIONS:
Behavioral: The cognitive rehabilitation program ReMind — Cognitive rehabilitation, i.e. psychoeducation, strategy training & retraining
  Other Names: ReMind-app

SUMMARY:
Many patients with primary brain tumors experience cognitive deficits and cognitive rehabilitation programs aim to alleviate these deficits.The cognitive rehabilitation program developed by the investigators proved effective in a large randomized controlled trial (RCT). To increase its accessibility, it was converted into the iPad-based cognitive rehabilitation program ReMind, which incorporates psychoeducation, strategy training and retraining. A pilot study and a randomized controlled trial are conducted, to evaluate the feasibility of the use of the program and the efficacy of the program in brain tumor patients after resective surgery.

DETAILED DESCRIPTION:
OBJECTIVE: To evaluate the immediate and longer-term effects of early cognitive telerehabilitation on cognitive performance and self-reported symptoms/functioning in patients with low-grade gliomas and meningiomas, in a prospective randomized trial.

HYPOTHESIS: Cognitive telerehabilitation after brain tumor surgery has both immediate and longer-term beneficiary effects on cognitive functioning and patient-reported outcomes.

STUDY DESIGN: In the first 6 months of the project a feasibility study will be conducted to ensure that adherence, patient experience, and potential attrition are acceptable.

Subsequently, a prospective randomized (waiting-list) controlled trial (RCT) will be performed. Information from the feasibility study will be used to modify the RCT when necessary. In the RCT, patients are randomized to early cognitive rehabilitation (3 months after surgery) or to a waiting-list control condition. The waiting-list control group will be offered the same cognitive rehabilitation program after they have undergone all study assessments. Assessment of cognitive performance and self-reported symptoms will be performed prior to surgery (T0), before cognitive rehabilitation (3 months after surgery, T3), immediately after cognitive rehabilitation (6 months after surgery, T6), and at half-year follow up (12 months after surgery, T12).

STUDY POPULATION/SAMPLE SIZE: Patients with presumed low-grade glioma or meningioma, who are scheduled for resective surgery, will be included in the study. Fifteen patients will be invited in feasibility study. Based on the yearly numbers of meningioma and low-grade glioma patients that are operated in the Elisabeth-TweeSteden Hospital Tilburg, it is expected that 60 patients will be randomized in the RCT per year for 2.5 years. With a maximum attrition rate of 33%, a minimum of 100 patients (50 per group) will be evaluated.

INTERVENTION: An evidence-based cognitive rehabilitation program that is provided via a tablet app. The program consists of retraining, and teaching and practicing of compensational strategies of attention, memory and executive functioning. Patients spend 3 hours per week during 2.5 month in this home-based program. They are monitored and supervised by a trainer.

OUTCOME MEASURES: Feasibility (accrual, attrition, adherence, patient experience) will be monitored in the feasibility study.

At several time points during the RCT, patients will be tested with the computerized test battery (for cognition; CNS VS), two additional cognitive tests and several self-report questionnaires. Testing is done prior to surgery, prior to cognitive rehabilitation (3 months), immediately after cognitive rehabilitation (6 months) and at half-year follow up (12 months post-surgery). Questionnaires on self-reported cognitive functioning, psychological symptoms (anxiety and depression), and fatigue will be administered on all assessments; the questionnaires on work status, professional functioning and community integration are administered at baseline and one-year follow-up only.

ELIGIBILITY:
Inclusion Criteria:

* The adult patient has a (supratentorial or infratentorial) brain tumor that is radiologically suspect for either a meningioma or low grade glioma
* The patient will undergo resective surgery for the brain tumor

Exclusion Criteria:

* tumor resection in the last year
* progressive neurological disease
* diagnose of (acute) psychiatric or neurological disorders in the last 2 years
* chemotherapy in the last 2 years
* Karnovsky Performance Scale under 70
* Surgery-related complication (morbidity or mortality e.g., thrombosis or heart attack)
* Lack of basic proficiency in Dutch
* IQ below 85, or (very) low cognitive skills
* Insufficient reading skills/visual impairment (limiting the ability to follow the cognitive rehabilitation program).
* Clinical referral to cognitive rehabilitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2015-07-01 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in objective cognitive functioning | 3, 6, and 12 months after surgery
  Objective cognitive functioning is measured with the computerized test battery CNS Vital Signs
Change in working memory | 3, 6, and 12 months after surgery
  Working memory is measured with the subtest Digit Span of the the Wechsler Adult Intelligence Scale (WAIS-III)
Change in word fluency | 3, 6, and 12 months after surgery
  Word fluency is measured with the Letter Fluency test

SECONDARY OUTCOMES:
Change in subjective cognitive functioning | 3, 6, and 12 months after surgery
  Subjective cognitive functioning is measured with the Cognitive Failures Questionnaire (CFQ)
Change in symptoms of fatigue | 3, 6, and 12 months after surgery
  Fatigue is measured with the Multidimensional Fatigue Inventory (MFI)
Change in symptoms of anxiety | 3, 6, and 12 months after surgery
  Anxiety is measured with the Hospital Anxiety and Depression Scale (HADS)
Change in symptoms of depression | 3, 6, and 12 months after surgery
  Depression is measured with the Hospital Anxiety and Depression Scale (HADS)
Change in subjective executive functioning | 3, 6, and 12 months after surgery
  Subjective executive functioning is measured with the Behavior Rating Inventory of Executive Function
Change in professional functioning (1) | One day before surgery vs. 12 months after surgery
  Professional functioning is measured with the Work Ability Index (WAI)
Change in professional functioning (2) | One day before surgery vs. 12 months after surgery
  Professional functioning is measured with the Work Limitation Questionnaire (WLQ)
Change in (social) participation | One day before surgery vs. 12 months after surgery
  Participation is measured with the Community Integration Questionnaire (CIQ)

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Erasmus Medical Center, Rotterdam
  - Medical Center Haaglanden, The Hague
  - Elisabeth-TweeSteden Hospital, Tilburg

IPD SHARING:
Plan to Share IPD: Undecided